CLINICAL TRIAL: NCT04693117
Title: Functional Impact of Interval Training on Muscle Mass and Strength in Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: REC/Lhr/338
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Obese; Muscle Strength; Interval Training
Keywords: Obesity; Body composition; Exercise testing
MeSH Terms: conditions — Obesity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): Participants were voluntarily participated by non-probability consecutive sampling. It was a one group study with a limitation of non-randomization. The interventional group had performed interval training for 12 weeks, 3 days/week (figure 1). They sedentary conferring to activity level (≥ 30-minute, 3 days/weeks, moderate-intensity physical activity). They were not participated in any interval training program before participating in the study from six months. Written consent was taken after demonstration of the purpose, procedure, and related pros and cons. They were instructed to participate regularly in interval training.
  Interventions: Other: Interval Training

INTERVENTIONS:
Other: Interval Training — All individual of interventional group participated in an interval training program, which comprised of 3 days/week for twelve weeks. A booklet was given to each participant containing instructions and guideline about interval training. The interval training program was introduced as prescribed previously.17 After the workout, a cool down period of 5 minutes was given during which they perform paddling with low speed. All training program was supervised by a qualified physical therapist.

SUMMARY:
The primary objective was to investigate the effectiveness of interval training and to evaluate the best available method for measuring body composition and functional capacity.

Thirty obese subjects consecutively voluntarily participated in the current study. They ranked sedentary according to their level of activity (≥ 30-minute moderate physical activity 3days/wk). The training sessions were divided into the warm-up phase, training phase and a cool-down phase. The training programs were completed 3days/week for 12 weeks. Body composition was calculated by skinfold thickness method and bio-impedance before and after training. Similarly, aerobic capacities were measured by lactate threshold testing and by Astrand submaximal testing.

ELIGIBILITY:
Inclusion Criteria:

* 30 obese (BMI ≥ 30) and
* Sedentary lifestyle subjects (sample size was calculated by using WHO sample size calculator)
* Age 30-45 years and
* Hypercholesteremia

Exclusion Criteria:

* hypertension,
* diabetes,
* cardiovascular diseases
* systemic diseases

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-12-28 (Actual)

PRIMARY OUTCOMES:
Anthropometric measurement (Body Mass Index) | 3 months
  Body Mass Index:
  BMI Weight Status Below 18.5 Underweight 18.5 - 24.9 Normal or Healthy Weight 25.0 - 29.9 Overweight 30.0 and Above Obese
Functional capacity | 3 Months
  The functional capacity was assessed by lactate threshold level and by Astrand submaximal testing by using standardized protocol.
  Lactate inflection point (LIP), is the exercise intensity at which the blood concentration of lactate and/or lactic acid begins to increase rapidly. It is often expressed as 85% of maximum heart rate or 75% of maximum oxygen intake.
Anthropometric measurement (Lean body mass) | 3 months
  Lean body mass:Lean body mass is calculated as the difference between total body weight and body fat weight, or more simply, the weight of everything except the fat. The range of lean body mass considered to be healthy is around 70% - 90% with women being towards the lower end of the range and men higher.
Functional Capacity | 3 months
  The functional capacity was assessed by Astrand submaximal testing by using standardized protocol.
  The Astrand Test is a submaximal cycle ergometer aerobic fitness test best suited in rehabilitation and health purposes. description: Athletes pedal on a cycle ergometer at a constant workload for 7 minutes. Heart rate is measured every minute, and the steady state heart rate is determined.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Shabbir, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sydo N, Abdelmoneim SS, Mulvagh SL, Merkely B, Gulati M, Allison TG. Relationship between exercise heart rate and age in men vs women. Mayo Clin Proc. 2014 Dec;89(12):1664-72. doi: 10.1016/j.mayocp.2014.08.018. Epub 2014 Oct 29. PMID 25441400
- [Background] Al-Shawwa B, Al-Huniti N, Titus G, Abu-Hasan M. Hypercholesterolemia is a potential risk factor for asthma. J Asthma. 2006 Apr;43(3):231-3. doi: 10.1080/02770900600567056. PMID 16754527
- [Background] Sobol NA, Hoffmann K, Frederiksen KS, Vogel A, Vestergaard K, Braendgaard H, Gottrup H, Lolk A, Wermuth L, Jakobsen S, Laugesen L, Gergelyffy R, Hogh P, Bjerregaard E, Siersma V, Andersen BB, Johannsen P, Waldemar G, Hasselbalch SG, Beyer N. Effect of aerobic exercise on physical performance in patients with Alzheimer's disease. Alzheimers Dement. 2016 Dec;12(12):1207-1215. doi: 10.1016/j.jalz.2016.05.004. Epub 2016 Jun 23. PMID 27344641
- [Background] Faude O, Kindermann W, Meyer T. Lactate threshold concepts: how valid are they? Sports Med. 2009;39(6):469-90. doi: 10.2165/00007256-200939060-00003. PMID 19453206
- [Background] Donges CE, Duffield R, Drinkwater EJ. Effects of resistance or aerobic exercise training on interleukin-6, C-reactive protein, and body composition. Med Sci Sports Exerc. 2010 Feb;42(2):304-13. doi: 10.1249/MSS.0b013e3181b117ca. PMID 20083961
- [Background] Kiss O, Sydo N, Vargha P, Edes E, Merkely G, Sydo T, Merkely B. Prevalence of physiological and pathological electrocardiographic findings in Hungarian athletes. Acta Physiol Hung. 2015 Jun;102(2):228-37. doi: 10.1556/036.102.2015.2.13. PMID 26100312